CLINICAL TRIAL: NCT06603701
Title: Follow up of Strength and Body Composition With Impedancemeter Device During the First 10 Days After Acute Stroke.
Brief Title: Sarcopenia in the Acute Stroke
Acronym: SARCOSTROKE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of the principal investigator
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUO-2023-10
Record Dates: First submitted 2024-08-16; First posted 2024-09-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Stroke, Acute
Keywords: Stroke; Body composition; Bioimpedancemetry; Sarcopenia
MeSH Terms: conditions — Stroke; Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Impedance measurement for acute stroke patient (Other): Acute stroke patients will benefit from impedance measurement and dynamometry to determine the evolution of sarcopenia rates.
  Interventions: Diagnostic Test: Bioimpedancemetry; Other: Dynamometry

INTERVENTIONS:
Diagnostic Test: Bioimpedancemetry — 2. Bioimpedancemetry at T1, T2, T3 ; the measurement will be
  1. Squeletic mass (total and for each of the 4 limbs)
  2. Angle phase (total and for each of the 4 limbs)
Other: Dynamometry — Dynamometry will be performed to assess the strength of each upper limb (deficient and non deficient) at T1, T2, T3

SUMMARY:
Regardless of the cause of immobilization, within days or weeks there is rapidly a decrease in strength and muscle mass, which can lead to sarcopenia. In severe strokes, immobilization and neurologic damage may be added to promote sarcopenia. Several studies in Asian populations confirm rapid increases in sarcopenia rates after stroke, but there are only rare data in Western populations. The aim of this work is to monitor during the first 10 days after a severe stroke leading to a reduction in ambulation, the evolution of muscle strength (studied in dynamometry), body composition (studied by impedance measurement) and sarcopenia rates. Investigators will also look for factors that predict the occurrence of this sarcopenia (such as sex, age, initial deficiency, stroke volume, swallowing disorders, etc.).

DETAILED DESCRIPTION:
In stroke patients, muscle damage combines many mechanisms such as immobilization, nutritional disorders , sympathetic activity, inflammation and denervation . These general factors explain that post-stroke sarcopenia is also observed on the side considered healthy .

Several meta-analyzes have been carried out on this subject . In the study by Inoue et al., which brings together 35 studies on the subject, the rates of sarcopenia observed were overall of the order of 15% before the stroke, of 30% in the 10 days post-stroke and of the order of 50% in the first semester . Only about 10 studies have been performed in the acute phase . However, the majority of these studies were performed in Asian populations (32 of them). But this is a population with demographic and physiological characteristics that are different from those in the West. Thus, body mass indices are lower and the representation of older people is higher in the population (the Japanese population is the oldest in the world).

Body composition may be a predictor of the course of recovery from stroke. In a cohort study it was thus shown by bioimpedance measurements that patients with the lowest muscle mass index had more severe neurological deficits at admission. They also had poorer functioning and longer hospital stays. Muscle mass is an independent variable in predicting what happens to people who have had a stroke.

Strokes cause motor deficits that reduce movement on the deficit side but also on the unaffected side. Sarcopenia (loss of strength and muscle mass) develops in the first few days after a stroke and worsens the consequences of neurologic damage. While immobilization rapidly leads to sarcopenia, sarcopenia has been poorly studied in acute stroke, especially in Asian populations, which are unrepresentative of Western populations.

The aims of this work are to:

1. Longitudinally determine rates of sarcopenia in the acute phase of stroke during follow-up over the first 10 days after stroke.
2. Determine the factors that predict the occurrence of sarcopenia (age, degree of initial deficiency, lesion volume, etc.)
3. Track body composition by segment (4 limbs and trunk) over time in impedance measurement, particularly by distinguishing between deficit and nondeficit. Investigators will distinguish the usual parameters (skeletal muscle mass, angle phase).
4. Monitor motor recovery of the deficient upper limb and determine whether muscle mass is a prognostic factor for recovery.

Measurement will be done at three time (T1, T2, T3) T1 corresponds to the first 72 hours post stroke T2 corresponds at 5 days (+/-1 days) T2 corresponds at 8 days (+/-1 days)

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke patient
* Over 18 years of age
* Functional Ambulation Categories (FAC) < 3
* NIHSS upper limb score ≥ 1
* Able to understand assessment instructions
* Non-objection to the study
* Affiliated with a social security scheme

Exclusion Criteria:

* Person under guardianship or curatorship.
* Person deprived of liberty
* Person under court protection
* Other neurological or rheumatological pathology limiting mobility
* Presence of a pacemaker or defibrillator.
* Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
rate of sarcopenia | Day 1
  The rate of sarcopenia will be defined using the maximum flexion force of the fingers measured on a digital Jamar dynamometer in the healthy upper limb.
rate of sarcopenia | Day 1
  The rate of sarcopenia will be define using appendicular muscle mass index (Kg/m2) measured by impedancemetry
rate of sarcopenia | Day 5
  The rate of sarcopenia will be defined using the maximum flexion force of the fingers measured on a digital Jamar dynamometer in the healthy upper limb.
rate of sarcopenia | Day 5
  The rate of sarcopenia will be define using appendicular muscle mass index (Kg/m2) measured by impedancemetry
rate of sarcopenia | Day 8
  The rate of sarcopenia will be defined using the maximum flexion force of the fingers measured on a digital Jamar dynamometer in the healthy upper limb.
rate of sarcopenia | Day 8
  The rate of sarcopenia will be define using appendicular muscle mass index (Kg/m2) measured by impedancemetry

SECONDARY OUTCOMES:
total skeletal muscle mass and per limb segment | Day 5
  total skeletal muscle mass and per limb segment (expressed in kg)
total skeletal muscle mass and per limb segment | Day 8
  total skeletal muscle mass and per limb segment (expressed in kg)
total angle phase and per limb segment | Day 5
  total angle phase and per limb segment expressed in degrees and evaluated at a frequency of 50kHz
total angle phase and per limb segment | Day 8
  total angle phase and per limb segment expressed in degrees and evaluated at a frequency of 50kHz
Muscular strength of the upper limb deficiency | Day 1
  Muscular strength of the upper limb deficiency expressed in Kg
Muscular strength of the upper limb deficiency | Day 5
  Muscular strength of the upper limb deficiency expressed in Kg
Muscular strength of the upper limb deficiency | Day 8
  Muscular strength of the upper limb deficiency expressed in Kg

CONTACTS AND LOCATIONS:
Overall Officials: Canan OZSANCAK, PH, Principal Investigator — CHU Orléans
Locations (1):
- CHU d'ORLEANS, Orléans, France

REFERENCES:
- [Background] Abe T, Iwata K, Yoshimura Y, Shinoda T, Inagaki Y, Ohya S, Yamada K, Oyanagi K, Maekawa Y, Honda A, Kohara N, Tsubaki A. Low Muscle Mass is Associated with Walking Function in Patients with Acute Ischemic Stroke. J Stroke Cerebrovasc Dis. 2020 Nov;29(11):105259. doi: 10.1016/j.jstrokecerebrovasdis.2020.105259. Epub 2020 Aug 28. PMID 33066891
- [Background] Herman SD, Friedman AC, Radecki PD, Caroline DF. Incidental prostatic carcinoma detected by MRI and diagnosed by MRI/CT-guided biopsy. AJR Am J Roentgenol. 1986 Feb;146(2):351-2. doi: 10.2214/ajr.146.2.351. No abstract available. PMID 3484585
- [Background] Arasaki K, Igarashi O, Ichikawa Y, Machida T, Shirozu I, Hyodo A, Ushijima R. Reduction in the motor unit number estimate (MUNE) after cerebral infarction. J Neurol Sci. 2006 Dec 1;250(1-2):27-32. doi: 10.1016/j.jns.2006.06.024. Epub 2006 Aug 9. PMID 16904126
- [Background] Arasaki K, Igarashi O, Machida T, Hyodo A, Ushijima R. Reduction in the motor unit number estimate (MUNE) after cerebral infarction. Suppl Clin Neurophysiol. 2009;60:189-95. doi: 10.1016/s1567-424x(08)00019-6. PMID 20715381
- [Background] Beckwee D, Cuypers L, Lefeber N, De Keersmaecker E, Scheys E, Van Hees W, Perkisas S, De Raedt S, Kerckhofs E, Bautmans I, Swinnen E. Skeletal Muscle Changes in the First Three Months of Stroke Recovery: A Systematic Review. J Rehabil Med. 2022 Oct 4;54:jrm00308. doi: 10.2340/jrm.v54.573. PMID 35848335
- [Background] Bellelli G, Zambon A, Volpato S, Abete P, Bianchi L, Bo M, Cherubini A, Corica F, Di Bari M, Maggio M, Manca GM, Rizzo MR, Rossi A, Landi F; GLISTEN Group Investigators. The association between delirium and sarcopenia in older adult patients admitted to acute geriatrics units: Results from the GLISTEN multicenter observational study. Clin Nutr. 2018 Oct;37(5):1498-1504. doi: 10.1016/j.clnu.2017.08.027. Epub 2017 Sep 5. PMID 28918171
- [Background] Bernhardt J, Hayward KS, Kwakkel G, Ward NS, Wolf SL, Borschmann K, Krakauer JW, Boyd LA, Carmichael ST, Corbett D, Cramer SC. Agreed Definitions and a Shared Vision for New Standards in Stroke Recovery Research: The Stroke Recovery and Rehabilitation Roundtable Taskforce. Neurorehabil Neural Repair. 2017 Sep;31(9):793-799. doi: 10.1177/1545968317732668. PMID 28934920